CLINICAL TRIAL: NCT05322460
Title: A Web-based Tailored Intervention to Improve the Quality of Life of Long-term Breast Cancer Survivors. A Randomized Controlled Trial
Brief Title: Web-based Intervention for Long-term Breast Cancer Survivors
Acronym: CUMACA-M
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cristina García-Vivar (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Cristina García-Vivar, Professor, Fundacion Miguel Servet
Organization: Fundacion Miguel Servet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPNA-CUMACA-B2022
Record Dates: First submitted 2022-03-28; First posted 2022-04-11 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Long-term Effects of Cancer Treatment; Long-term Effects Secondary to Cancer Therapy in Adults
Keywords: Cancer survivors; Long-Term Cancer Survivors; Long Term Cancer Survivors; Survivorship

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The CUMACA-M Program will focus on a web-based tailored intervention, using artificial intelligence, for Long-Term Survivors of Breast Cancer. It will be structured into modules related to the specific needs of LS-BS, including physical, psychological, and social needs
  Interventions: Other: CUMACA-M Program
- Control group (No Intervention): Usual care in the nursing consultation in primary care

INTERVENTIONS:
Other: CUMACA-M Program — The CUMACA-M Program will focus on a web-based tailored intervention, using artificial intelligence, for Long-Term Survivors of Breast Cancer. It will be structured into modules related to the specific needs of LS-BS, including physical, psychological, and social needs
  Arms: Intervention group

SUMMARY:
The number of breast cancer survivors is growing. More cured women are becoming long-term survivors of breast cancer (LS-BC) at least 5 years after diagnosis and after treatment has been completed. Some of these LS-BC return to daily life without any problems; however, in many cases, they experience and have to deal with physical sequelae (chronic fatigue, pain, etc.) psychological sequelae (anxiety, depression, fear of recurrence, etc.) and social sequelae (altered interpersonal relationships, difficulty in returning to work, etc.). For many LS-BC, these health problems are not being met by health professionals. Thus there is a need to promote greater continuity and coordination between specialized oncology care and primary health care in order to enhance specific follow-up of these women in the community. However, the role of the primary health care team in the provision of care in the long-term cancer survival is not clearly defined and few actions have been aimed at improving care activities, standardizing procedures and protocols, developing documentation and registries and updating the training of health care professionals. Therefore, this study aim to design, implement, and evaluate a web based tailored intervention, using artificial intelligence, to improve the quality of life of long-term breast cancer survivors, and self-efficacy for the management of late sequelae from primary care.

DETAILED DESCRIPTION:
Hypothesis: A web-based tailored intervention, based on the prevention and management of physical and psychosocial late effects due to cancer treatment and aimed at improving the coexistence of long-term breast cancer, will be more effective in improving quality of life and self-efficacy for the management of late sequelae from Primary Care, than conventional care offered in Primary Care. Aim: To design, implement and evaluate the effectiveness of a web-based tailored intervention, based on artificial intelligence, to improve the quality of life of long-term survivors of breast cancer and self-efficacy for the management of late sequelae from Primary Healthcare. Methodology: Randomized controlled trial (following the Medical Research Council methodological framework). Phase I. Design of a personalized digital intervention based on the results of a review of the available evidence on the needs of long-term survivors (LS-BC) of breast cancer and agreed with a panel of experts. It will be designed in web/mobile application format. The use of algorithms will allow the personalization of the contents according to the needs. Phase II. Piloting: Pre-experimental design pretest-postest with one group, by means of a convenience sampling with LS-BC women, who meet the selection criteria. The collection of sociodemographic and clinical data, as well as the variables under study; quality of life (QOL-BC), self-efficacy in the management of cancer sequelae (Self-Efficacy for Managing Chronic Disease). The participants will use a web application and will test the usability and functionality. Phase III. Implementation of the intervention: Randomized controlled trial. Random sampling of LS-BC and random assignment to the intervention group (CUMACA-M program) or control group (standard care). A protocol will be designed that allows the collection of data and variables (Phase II) and satisfaction with the intervention (CSQ-8), at pre-intervention, and at 3, 6 and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with breast cancer
* having completed active oncological treatments (chemotherapy and/or radiotherapy) in a period of time greater than five years,
* be free of disease at the time of data collection
* be a woman and over 18 years of age
* have knowledge of Internet use.

Exclusion Criteria:

* Women with a diagnosis of cancer other than breast cancer
* Recurrence of cancer or metastasis that causes a new treatment
* Being in active treatment for recurrence or new cancer
* Being a man

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Quality of life Cancer Survivor (QOL-CS) | Changes from baseline, 3-months, 6 months, and 9 month
  The QOL-CS, Spanish version (Ferrell B, Hassey-Dow K, Grant M. Quality of Life Patient/Cancer Survivor Version (QOL-CS) [Internet]. Measurement Instrument Database for the Social Science. 2012). Scale specific for cancer survivor. Likert-type scale with 10 options (1 extremely poor and 10 excellent) with 41 items that measure the four domains of quality of life: physical, psychological, social and spiritual well-being.
Self-Efficacy for Managing Chronic Disease | Changes from baseline, 3-months, 6 months, and 9 month
  The Self-Efficacy for Managing Chronic Disease- 6-Item Scale (SEMCD-6) (Ritter PL, Lorig K. The English and Spanish Self-Efficacy to Manage Chronic Disease Scale measures were validated using multiple studies. J Clin Epidemiol. 2014; 67(11): 1265-73). The scale is structured in 6 items related to symptom control, role performance, emotional state and communication with health professionals
Sociodemographic data of LS-BC | Baseline
  Sociodemographic data of the LS-BC (age, sex, marital status, educational level, employment status) will be collected by means of an ad hoc questionnaire at the beginning of the intervention.

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | 4 weeks
  The satisfaction with the CUMACA-M Program will be measured using the Spanish version of the Client Satisfaction Questionnaire (CSQ-8) (Attkisson CC, Greenfield TK. The UCSF Client Satisfaction Scales: I. The Client Satisfaction Questionnaire-8. In Maruish M (Ed). 2004). This scale is structured into 8 items with has five response options (from very dissatisfied to very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Garcia Vivar, PhD, Principal Investigator — Universidad Pública de Navarra
Locations (1):
- Public University of Navarre, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pimentel-Parra GA, Soto-Ruiz N, Escalada-Hernandez P, San Martin-Rodriguez L, Garcia-Vivar C. EHealth intervention for quality of life in long-term breast cancer survivors: Randomized controlled trial. J Natl Cancer Inst. 2026 Jan 24:djag020. doi: 10.1093/jnci/djag020. Online ahead of print. PMID 41581214